CLINICAL TRIAL: NCT05469516
Title: Superficial MFU-V and Diluted Calcium Hydroxyapatite for the Improvement of Lower Face Skin Quality and Wrinkles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cutis Medical Laser Clinics Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Cutis
Record Dates: First submitted 2022-06-03; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: This is a single centre prospective pilot study to evaluate the efficacy of combining MFU-V and diluted CaHA for improving skin quality on the lower face.
  Treatment protocols are as follows:
  1. MFU-V delivered to the lower face areas as drawn using a single transducer with a focal depth of 1.5mm (following a previously published paper (Lowe, 2021) but with extension of the lower treatment area to the two-ruler width (Ulthera marking ruler) as treatment zones. Application will be delivered through a cross-hatching technique.
  2. Immediately following MFU-V or up to a week after, diluted CaHA will be administered following the Global Consensus Guidelines published in 2018 by de Almeida et al as follows 1) 1 syringe or 1.5ml of CaHA diluted 1:1 with saline for a total of 3ml of solution or 1.5 diluted CaHA per side will be injected in the subdermal plane with a cannula using a retrograde fanning technique.
Masking Description: • Blinded assessment of aesthetic improvement at each visit as follows: Blinded reviewer to make qualitative comparisons of images of treated arms vs. baseline at each follow-up visit. If the reviewer perceived an improvement, he/she ask will be asked to select the correct post-treatment photograph
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Ultherapy and Radiesse (Experimental): Delivered to the lower face areas as drawn using a single transducer with a focal depth of 1.5mm (following a previously published paper (Lowe, 2021) but with extension of the lower treatment area to the two-ruler width (Ulthera marking ruler) as treatment zones. Application will be delivered through a cross-hatching technique.
  Immediately following MFU-V or up to a week after, diluted CaHA will be administered following the Global Consensus Guidelines published in 2018 by de Almeida et al as follows 1) 1 syringe or 1.5ml of CaHA diluted 1:1 with saline for a total of 3ml of solution or 1.5 diluted CaHA per side will be injected in the subdermal plane with a cannula using a retrograde fanning technique.
  Interventions: Device: Ulthera System [Ulthera, Inc.]; Device: Merz Radiesse Injectable Implant

INTERVENTIONS:
Device: Ulthera System [Ulthera, Inc.] — The Ulthera System is indicated for: - Use for noninvasive dermatological sculpting and lifting of the dermis: Upper Face, Lower Face, Neck, Décolletage.
  - Non-invasive treatment of Axillary Hyperhidrosis
Device: Merz Radiesse Injectable Implant — Radiesse injectable implant is an opaque, sterile, non-pyrogenic, semi-solid, cohesive implant. The principal component is synthetic CaHA suspended in a gel carrier that consists primarily of water (sterile water for injection, United States pharmacopeia (USP)), glycerin (USP), and sodium carboxymethylcellulose (USP). Radiesse injectable implant (1.5mL syringe unit) has a CaHA particle size range of 25-45 microns and should be injected sub-dermally with a 27 gauge needle.

SUMMARY:
Aging, genetics and environmental factors contribute to multiple changes on the surface of the skin. These present with pigmentation, volume loss, loss of elasticity and loss of collagen. Altogether, areas of the face becomes "crepey", with resulting rhytids and an obvious appearance of thin and fragile skin. These are typically dermal manifestations of elastin and collagen loss resulting in a collective term of loss of "skin quality".

Current treatments to improve these changes involve the use of skincare, chemical peels, as well as more invasive repeated treatments such as microneedling and laser resurfacing. These commonly require repeated treatments and several days of downtime. More recently, treatment with a hybrid preparation of high and low-molecular weight complexes that are thermally cross-linked (Profhilo) has been suggested to stimulate collagen and elastin formation, thereby resulting in improvement in skin quality.

DETAILED DESCRIPTION:
Aging, genetics and environmental factors contribute to multiple changes on the surface of the skin. These present with pigmentation, volume loss, loss of elasticity and loss of collagen. Altogether, areas of the face becomes "crepey", with resulting rhytids and an obvious appearance of thin and fragile skin. These are typically dermal manifestations of elastin and collagen loss resulting in a collective term of loss of "skin quality".

Current treatments to improve these changes involve the use of skincare, chemical peels, as well as more invasive repeated treatments such as microneedling and laser resurfacing. These commonly require repeated treatments and several days of downtime. More recently, treatment with a hybrid preparation of high and low-molecular weight complexes that are thermally cross-linked (Profhilo) has been suggested to stimulate collagen and elastin formation, thereby resulting in improvement in skin quality However, the evidence for this remains limited. Microfocused Ultrasound with Visualization (MFU-V) and Calcium hydroxylapatite (CaHA) have each been unequivocally proven to stimulate neocollagenesis and elastogenesis, leading to improvement in skin laxity. A recent study of a single-treatment single-depth of superficial MFU-V was found to result in aesthetic improvement of the accordion lines. In addition, there is recent evidence that CaHA in a hyperdiluted form can stimulate collagen and elastin formation. Indeed, this group of investigators has recently published the effectiveness of a single treatment of a combination MFU-V and diluted CaHA for improving brachial skin laxity. Arguably, there is a need to publish additional studies on these interventions for improving firmness and skin quality. In addition, there may be a theoretical cumulative benefit in using both treatments for improving skin quality, although the effectiveness of this combination has not been demonstrated.

With this background, the main rationale of performing this study is to demonstrate the safety and efficacy of a multimodality approach with a single treatment of superficial MFU-V and diluted CaHA for improvement of skin quality in Asian and Caucasian patients. The investigators selected Lower Face as the target area for the following reasons: 1) The Lower Face manifests the greatest with thinning, fine wrinkling and general fragility of the skin, 2) Volumization is not always aesthetically pleasing in this area but firmness of the skin is, 3) This area is an established treatment area for MFU-V, CaHA but not with other treatment options such as Profhilo.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with lower face wrinkles
* Otherwise generally healthy.
* Physically and mentally capable to provide informed consent to the study.
* Agreement to attend all follow-up visits as scheduled

Exclusion Criteria:

* Pregnancy or lactation;
* History of allergic reaction to calcium hydroxylapatite injection;
* Active local infections or skin diseases that might alter wound healing
* Acne or keloidal scarring
* Use of immunosuppressive drugs
* Any other diseases which can affect the wound-healing process
* Any procedures affecting facial wrinkles or skin quality in the lower face for the duration of the study
* Microdermabrasion and Peels
* Acne treatments
* Filler and Botulinum Toxin treatments
* Radiofrequency, Laser, IPL, Ultrasound
* Patients that had cosmetic treatments within 3 months of the baseline visit in the treatment area
* Subjects with dermatologic conditions in the treatment area including:
* Acne
* Rosacea
* Eczema
* Psoriasis
* Actinic keratosis,
* Severe sun damage
* Scars or a history of keloids

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in Skin Quality | 1 Month, 3 Months and 6 Months post intervention
  Pre and post treatment comparison of change in skin quality. These will be measured using Quantificare LifeViz Micro, an established tool to objectively measure and validate treatment results of skin quality which will allow to accurately quantify changes with specific measurement tools.
Change in Wrinkle Reduction | 1 Month, 3 Months and 6 Months post intervention
  Pre and post treatment comparison of change in dimensions of fine lines (volume/depth/length). These will be measured using Quantificare LifeViz Micro, an established tool to objectively measure and validate treatment results of lines, which will allow to accurately quantify changes with specific measurement tools.

SECONDARY OUTCOMES:
Visual Aesthetic Improvement Score | 1 Month, 3 Months and 6 Months post intervention
  Pre and post treatment comparison of Visual Aesthetic Improvement Score of standardized patient photographs by study investigators. Both VISIA Imaging photographs and standard photographs will be used.

OTHER OUTCOMES:
Patient Satisfaction | 1 Month, 3 Months and 6 Months post intervention
  To evaluate patient satisfaction of change of lower face skin quality using a 5 point scale where 1 means strongly disagree and 5 means strongly agree.
Establish Number of Adverse Events | 1 Month, 3 Months and 6 Months post intervention
  Count the number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Cutis Medical Laser Clinics, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

REFERENCES:
- [Background] Narins RS, Carruthers J, Flynn TC, Geister TL, Gortelmeyer R, Hardas B, Himmrich S, Jones D, Kerscher M, de Maio M, Mohrmann C, Pooth R, Rzany B, Sattler G, Buchner L, Benter U, Breitscheidel L, Carruthers A. Validated assessment scales for the lower face. Dermatol Surg. 2012 Feb;38(2 Spec No.):333-42. doi: 10.1111/j.1524-4725.2011.02247.x. PMID 22316189
- [Background] Shoshani D, Markovitz E, Monstrey SJ, Narins DJ. The modified Fitzpatrick Wrinkle Scale: a clinical validated measurement tool for nasolabial wrinkle severity assessment. Dermatol Surg. 2008 Jun;34 Suppl 1:S85-91; discussion S91. doi: 10.1111/j.1524-4725.2008.34248.x. PMID 18547187
- [Background] Information and Instruction Manual for Cutometer® dual MPA 580. English 2019/02 DK. [Available from: https://www.courage-khazaka.de/en/16-wissenschaftliche-produkte/alle-produkte/178-cutometer-e
- [Result] Lowe S. Single Treatment, Single Depth Superficial Microfocused Ultrasound with Visualization for Rhytid Improvement. Plast Reconstr Surg Glob Open. 2021 Jul 13;9(7):e3662. doi: 10.1097/GOX.0000000000003662. eCollection 2021 Jul. PMID 34277316
- [Result] Ramirez S, Puah IBK. Effectiveness of combined microfocused ultrasound with visualization and subdermal calcium hydroxyapatite injections for the management of brachial skin laxity. J Cosmet Dermatol. 2021 Dec;20(12):3871-3879. doi: 10.1111/jocd.14573. Epub 2021 Oct 29. PMID 34716645
- [Result] Goldie K, Peeters W, Alghoul M, Butterwick K, Casabona G, Chao YYY, Costa J, Eviatar J, Fabi SG, Lupo M, Sattler G, Waldorf H, Yutskovskaya Y, Lorenc P. Global Consensus Guidelines for the Injection of Diluted and Hyperdiluted Calcium Hydroxylapatite for Skin Tightening. Dermatol Surg. 2018 Nov;44 Suppl 1:S32-S41. doi: 10.1097/DSS.0000000000001685. PMID 30358631
- [Result] de Almeida AT, Figueredo V, da Cunha ALG, Casabona G, Costa de Faria JR, Alves EV, Sato M, Branco A, Guarnieri C, Palermo E. Consensus Recommendations for the Use of Hyperdiluted Calcium Hydroxyapatite (Radiesse) as a Face and Body Biostimulatory Agent. Plast Reconstr Surg Glob Open. 2019 Mar 14;7(3):e2160. doi: 10.1097/GOX.0000000000002160. eCollection 2019 Mar. PMID 31044123
- [Result] Casabona G, Michalany N. Microfocused ultrasound with visualization and fillers for increased neocollagenesis: clinical and histological evaluation. Dermatol Surg. 2014 Dec;40 Suppl 12:S194-8. doi: 10.1097/DSS.0000000000000231. No abstract available. PMID 25417575